CLINICAL TRIAL: NCT02599103
Title: The Effects of Various Cooking Oils on Health Related Biomarkers in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academia Sinica, Taiwan (Other)
Responsible Party: Principal Investigator, Wen-Harn Pan, Institute of Biomedical Sciences, Academia Sinica, Taiwan
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AS-IRB02-102083
Record Dates: First submitted 2015-09-15; First posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Olive Oil; Soybean Oil; Palm Oil; tallow

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- fat-free milkshake (Placebo Comparator)
  Interventions: Other: Fat-free milkshake
- Olive oil (Active Comparator)
  Interventions: Other: Olive oil
- soybean oil (Experimental)
  Interventions: Other: Soybean oil
- fried soybean oil (Experimental)
  Interventions: Other: Fried soybean oil
- palm oil (Experimental)
  Interventions: Other: Palm oil
- fried palm oil (Experimental)
  Interventions: Other: Fried palm oil
- camellia oil (Experimental)
  Interventions: Other: Camellia oil
- fried camellia oil (Experimental)
  Interventions: Other: Fried camellia oil
- tallow (Experimental)
  Interventions: Other: Tallow
- fried tallow (Experimental)
  Interventions: Other: Fried tallow

INTERVENTIONS:
Other: Fat-free milkshake — participants drinks a fat-free milk shakes
  Arms: fat-free milkshake
Other: Olive oil — participants drinks the milk shakes prepared from 60g of olive oil
  Arms: Olive oil
Other: Soybean oil — participants drinks the milk shakes prepared from 60g of soybean oil
  Arms: soybean oil
Other: Fried soybean oil — participants drinks the milk shakes prepared from 60g of fried soybean oil
  Arms: fried soybean oil
Other: Palm oil — participants drinks the milk shakes prepared from 60g of palm oil
  Arms: palm oil
Other: Fried palm oil — participants drinks the milk shakes prepared from 60g of fried palm oil
  Arms: fried palm oil
Other: Camellia oil — participants drinks the milk shakes prepared from 60g of camellia oil
  Arms: camellia oil
Other: Fried camellia oil — participants drinks the milk shakes prepared from 60g of fried camellia oil
  Arms: fried camellia oil
Other: Tallow — participants drinks the milk shakes prepared from 60g of tallow
  Arms: tallow
Other: Fried tallow — participants drinks the milk shakes prepared from 60g of fried tallow
  Arms: fried tallow

SUMMARY:
Fats and oils play important roles in maintaining human nutrition and health through providing energy, essential fatty acids, and acting as modulators of many biological processes (signal transduction, immunity and inflammation). Due to differences in the fatty acid composition and content of antioxidants of individual cooking oils, the degree of oxidative and thermolytic reactions may vary oil by oil. It is lack of human feeding study to investigate the molecular mechanisms on how and which deep-fried oil exerts its adverse effects. The investigators are also lack of biomarkers for monitoring deep-fried oil exposure. Therefore, the purpose of this study is to compare how human body responds differently to several popular uncooked and deep-fried oils with varied fatty acid compositions with respect of oxylipin profile, inflammatory markers, non-targeted metabolomics, and transcriptomics. The investigators will recruit 20 volunteers, provided them once a week the milk shakes prepared from 60g of olive oil, soybean oil, palm oil, camellia oil, tallow (butter), and deep-fried oils of the last 4, respectively; in comparison with a no-fat milk shake control. The experiments lasted for 10 weeks.。Each time; serum, plasma, whole blood and urine samples were collected at baseline, after 2 hours, and after 4 hours. The investigators anticipate to find biomarker(s) for deep-frying, and contribute to the understanding of molecular mechanisms on how deep-fried oils exert adverse effects toward health through integrative omics or so-called system biology approaches.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, non-drinker, usual dietary intake
* BMI : 18.5~27 kg/m2

Exclusion Criteria:

1. Over the past two weeks have suffered from acute illness.
2. None of the subjects was taking any supplemental vitamins, antioxidants or medication at that time.
3. Taking steroids or non-steroidal anti-inflammatory drug, such as Aspirin or Panadol in the past one week.
4. Cancer or other severe diseases was diagnosed.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The changs of metabolomics profile between before and after oil consumption | baseline to 2 hours and 4 hours after oil consumption
  This is a metabolomics study. We measured retention time (min), mass and abundance of serum metabolites with LC-QTOF at 3 time points. Then, we compared the abundance of metabolites between different oil consumption time ( before and after ) and assessed the health effects of cooking oils.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, Ph.D., Principal Investigator — Institute of Biomedical Sciences, Academia Sinica